CLINICAL TRIAL: NCT06864325
Title: Assessment of Changes in Functional Status and Quality of Life in Seniors Engaging in Virtual Reality-based Physical Activity: Influence of Diet, Oral Microflora Composition, Blood Morphology, and Anthropometric Parameters
Brief Title: VR Gaming and Its Impact on Functional Status and Quality of Life in Seniors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Opole University of Technology (Other)
Responsible Party: Principal Investigator, Żaneta Grzywacz, Principal Investigator, The Opole University of Technology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OpoleUofTech5
Record Dates: First submitted 2025-02-24; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Older Adults
Keywords: virtual reality; functional statut; quality of life; older adults

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR group (Experimental): The VR group underwent a four-week training program, with sessions held three times per week, each lasting 20 minutes. Initially, an introductory session was organized to familiarize the participants with virtual reality. Following this, the structured training program consisted of 12 sessions over the four-week period. All sessions were conducted in a seated position to ensure comfort and safety.
  Interventions: Other: VR-training
- Control group (No Intervention): The control group was a passive group that do not receive any specific intervention, engaging only in the standard daily exercises provided at the nursing home.

INTERVENTIONS:
Other: VR-training — The VR gaming experience is based on the commercial rhythm game Beat Saber, featuring songs by Queen with varying rhythms and tempos. Players receive visual stimuli in the form of colored square blocks and must slice them in time with the music using the corresponding right or left hand. The blocks must be cut with a lightsaber of the same color. To ensure the safety of older adults, heart rate and energy expenditure were monitored throughout each session, while oxygen saturation was assessed before and after the exercises. Participants playe the game in comfortable conditions: the game loaded directly into the headset and VR glasses synchronized with portable screens to allow monitoring and assistance if needed. Before each session, the headset was adjusted to fit the participant's head dimensions, and corrective glasses were provided if required. The VR setup included a Meta Quest 2 headset with goggles and user-friendly controllers equipped with sensors (Meta Platforms, U.S.).
  Other Names: VR-gaming
  Arms: VR group

SUMMARY:
This project examined the impact of virtual reality (VR)-based physical activity on the functional status and quality of life (QoL) of older residents in a nursing home. It is know that VR-related therapy and activation programs help in a positive attitude toward health and emotions, reduce susceptibility to depression and social isolation, and enhance engagement in physical activities. As an atrractive and motivating tools, VR have the potential to promote greater physical activity and overall improvement, including functional status and QoL in older adults. Such findings indicate that incorporating VR into exercise programs for the older adults may enhancements in functional status and QoL compared to traditional, non-VR-based therapy.

The primary goal of this study was to assess changes in functional status and QoL in older participants in VR-based physical activity. The project involves a comprehensive evaluation, including assessments of physical and psychomotor fitness, body composition, key blood morphology parameters, lipid profile, blood glucose levels, oral microbiome composition, and overall well-being. Additionally, psychological factors such as anxiety levels is examined, assuming that these parameters may improve through VR-enhanced physical activity.

The investigators hypothesize that VR-based therapy will leads to significant improvements in psychomotor and functional fitness, exercise tolerance, and overall well-being, thereby enhancing the QoL in older adults. The findings of this research may contribute to the development of innovative programs aimed at supporting elderly individuals in maintaining and improving their functional status-whether during recovery, rehabilitation, or in sustaining optimal physical and mental health.

DETAILED DESCRIPTION:
The project involved older adults residing in a nursing home, who are randomly assigned to one of two study groups: the intervention group with participants undergo virtual reality (VR)-based training, and the control group with participants engage in standard activities provided by the nursing home. Our study design assumes that the participants will undergo 2 rounds of testing conducted before therapy to evaluate the subjects' initial condition (T0 testing), and after therapy to assess the effects of the intervention (T1 testing). These assessments will be separated by a four-week period during which the intervention group completes 12 VR-based sessions.

Scope of assessments at T0 and T1 includes:

I. survey studies - introductory custom questionnaire, questionnaires assessing mental health, quality of life, functional fitness in daily activities, complex activities of daily living, and functional independence; II. psychomotor assessments - tests of eye-hand coordination and attention concentration; III. physical fitness assessment - grip strength measurements, general physical fitness evaluation, analysis of body composition; IV. lifestyle and biological assessments - oral microbiota assessment, laboratory tests including peripheral blood morphology, lipid profile, glucose level and C-reactive protein concentration, and analysis of nutritional habits.

Moreover, participants in the intervention group during VR gaming possess evaluation of parameters indicating intervention effectiveness, and measurement of heart rate, energy expenditure, and oxygen saturation levels.

ELIGIBILITY:
Inclusion criteria:

* age 60 or older
* signing an informed consent to participate in the study
* willingness to participate in the therapy program.

Exclusion criteria:

* lack of consent
* contraindications to VR headset using (current temporary conditions: fatigue or exhaustion, drowsiness, nausea, anxiety or stress, cold, flu)
* chronic conditions (cancer in an intensive treatment phase, inability to exercise, visual or auditory disorders preventing VR goggles use, cognitive disorders that hindered understanding exercise instructions or cooperation with the researcher).

Eligibility was determined by a physician who assessed each participant's health condition, and screened for contraindications to a head-mounted display VR use.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2024-07-17 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Own survey research | 76 days
  The study included a custom questionnaire assessing demographic data, physical activity, quality of life, diet, oral prophylaxis, existing diseases, and medications taken, administered before intervention (at the T0). A follow-up questionnaire evaluated participants' impressions of the VR intervention is conducted after intervention (T1).
Survey research - the levels of anxiety and depression | 76 days
  At both T0 and T1 time points mental health was assessed using the Hospital Anxiety and Depression Scale (HADS).
Survey research - quality of life | 76 days
  At both T0 and T1 time points quality of life was measured with the World Health Organization's short Quality of Life Scale (WHOQOL-BRIEF)
Survey research - functional ability | 76 days
  At both T0 and T1 time points a functional ability in daily life was assessed through Activities of Daily Living (ADL) according to the Katz Index.
Survey research - activities of daily living | 76 days
  At both T0 and T1 time points Instrumental Activities of Daily Living (IADL) using the Lawton Scale.
Survey research - functional independence | 76 days
  At both T0 and T1 time points a functional independence was measured with the Functional Independence Measure (FIM).
Psychomotor assessments - tests of eye-hand coordination (EHC) and attention concentration (AC), | 76 days
  The cross visual motor test using the Piórkowski apparatus (PIOR/ATB 2.0) was used to assess EHC and AC. During the test, the participant was seated comfortably in front of the apparatus with their hands positioned over the buttons. The following test pattern was used: a duration of 90 seconds, with 1-second light intervals and stimulus frequency of 90 stimuli per 90 seconds. On the device's panel, lights were illuminated in random sequences, and the participant had to respond immediately by pressing the corresponding button as quickly and accurately as possible. The device recorded the subject's movements, reaction times and errors for each light stimulus. The test was conducted over three consecutive trials and an average score was calculated for each metric.
Physical fitness assessment - grip strength measurements | 76 days
  The test was conducted in a sitting position with the forearm resting on a table and the elbow bent at a 90-degree angle, The participant clenched their hand for 3 seconds; the test was repeated 3 times. The average result was then compared to normative values for muscle strength
Physical fitness assessment - upper body strength | 76 days
  The assessment was conducted using a Arm Curl Test - a part of Fullerton Functional Fitness Test. The participant sits on a chair, holding a weight (approximately 2.27 kg for women and 3.63 kg for men) in the dominant hand. The arm was positioned downward alongside the chair, perpendicular to the floor, with the palm facing inward. Upon the "start" signal, the participant bends the elbow, lifting the weight toward the shoulder, and then returns to the starting position. The total number of correctly performed repetitions within 30 seconds was recorded.
Physical fitness assessment - shoulder flexibility | 76 days
  The assessment was conducted using a Back Scratch Test - a part of the Fullerton Functional Fitness Test. Performed in a standing position. The participant attempted to touch the middle fingers of both hands behind the back using a 30 cm ruler. One arm was positioned over the shoulder, reaching down the middle of the back with the elbow pointing outward, while the other arm reaches up from below. The distance between the fingertips was measured to assess flexibility.
Physical fitness assessment - lower body strength | 76 days
  The assessment was conducted using Chair Stand Test - a part of the Fullerton Functional Fitness Test. The participant sited on a chair with arms crossed over the chest. Upon the "start" signal, they stand up fully and then sit back down. The number of complete stands performed within 30 seconds was recorded.
Physical fitness assessment - lower body flexibility | 76 days
  The assessment was conducted using Chair Sit-and-Reach Test - a part of the Fullerton Functional Fitness Test. While sitting on the edge of a chair, the participant extended one leg straight forward with the heel resting on the floor. Keeping the back straight and arms extended toward the toes, they lean forward as far as possible, attempting to reach their toes. The distance between the fingertips and toes was measured to assess lower body flexibility.
Physical fitness assessment - speed, agility, and balance | 76 days
  The assessment was conducted using 8-Foot Up-and-Go Test - a part of the Fullerton Functional Fitness Test. The participant started seated in a chair. Upon the "start" signal, they stand up, walk as quickly as possible to a marker placed 2.44 meters (8 feet) away, turn around, return to the chair, and sit down. The time taken to complete the task was recorded, assessing agility and dynamic balance.
Physical fitness assessment - aerobic endurance | 76 days
  The assessment was conducted using 2-Minute Step Test - a part of the Fullerton Functional Fitness Test. The participant marched in place for two minutes, lifting their knees to a height midway between the kneecap and hip. The number of times the right knee was raised is counted, providing an estimate of aerobic endurance.
Lifestyle and biological assessments - oral microbiota | 76 days
  For assess oral microbiota, the oral swabs were collected by qualified medical personnel. Biochemical identification of bacterial species present in the oral cavity, including Prevotella intermedia, Porphyromonas gingivalis, Fusobacterium nucleatum, Leptotrichia buccalis, and Propionibacterium ssp., were conducted using API biochemical strip tests.
Lifestyle and biological assessments - laboratory tests | 76 days
  The laboratory tests included blood morphology and biochemical analysis (lipid profile, glucose level and C-reactive protein concentration). The assessment were conducted using standard analyses in the diagnostic laboratory.
Lifestyle and biological assessments - adherence to healthy eating principles | 76 days
  The adherence to healthy eating principles was performed via nursing home menus evaluation and using the Healthy Diet Index (HDI). HDI was expressed in point scale.
Lifestyle and biological assessments - compliance with dietary recommendations | 76 days
  The compliance with dietary recommendations was performed via nursing home menus evaluation and using the Healthy Eating Index (HEI). HEI was expressed in point scale.
Lifestyle and biological assessments - quantitative diet analysis | 76 days
  A quantitative diet evaluation determined nutrient content, including protein, fat, carbohydrates, fiber, vitamins, and minerals. The analysis was performed via nursing home menus evaluation. The diet was assessed according to nutritional standards for the older adults.
Lifestyle and biological assessments - qualitative diet assessment | 76 days
  A qualitative assessment was performed via nursing menus evaluation analysis and using Food Quality Index (DQI), Starzyńska-Bielińska test, Szewczyński's classification, and Block's questionnaire. The results were expressed in point scales.
Anthropometric data - height | 76 days
  Height was measured using a heightmeter in centimeters.
Anthropometric data - weight | 76 days
  Weight was carried out using the InBody 120 analyzer. Body weight was measured in kg.
Anthropometric data - body mass index | 76 days
  Weight and height were combined to report body mass index (BMI). BMI was expressed in kg/m^2
Physical fitness assessment - body composition analysis | 76 days
  Body composition was carried out using the InBody 120 analyzer, which utilizes bioelectrical impedance analysis. This method enables an objective evaluation of muscle mass, body fat percentage, body mass index, stored energy, and water content in the body.
Anthropometric data - body circumferences | 76 days
  Waist and hip circumference were measured using an electronic measuring tape in centimeters.
Anthropometric data - skinfold thickness | 76 days
  Skinfold thickness was measured using a professional caliper.

SECONDARY OUTCOMES:
Heart ratio | 76 days
  To ensure the safety of older adults, heart ratio was monitored throughout each session of VR-based training. Data were collected using fitness trackers, specifically the Fitbit Charge 6, known for its accuracy in data collection during moderate physical activity.
Energy expenditure | 76 days
  To ensure the safety of older adults, energy expenditure was monitored throughout each session of VR-based training. Data were collected using fitness trackers, specifically the Fitbit Charge 6, known for its accuracy in data collection during moderate physical activity.
Saturation | 76 days
  To ensure the safety of the elderly, saturation was monitored during each VR-based training session. Data were collected using a fingertip pulse oximeter

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Faculty of Physical Education and Physiotherapy, Opole University of Technology, Opole
  - Faculty of Production Engineering and Logistics, Opole University of Technology, Opole

IPD SHARING:
Plan to Share IPD: Yes
It was decided to provide free access to the analysed data. The data will be available upon request sent to PI: z.grzywacz@po.edu.pl
Supporting Information: Study Protocol
Time Frame: 6 months
Access Criteria: The data will be available upon request sent to PI